CLINICAL TRIAL: NCT06974799
Title: Evaluation of Metabolomic Biomarkers in Pulmonary Fibrosis
Brief Title: Metabolomic Biomarkers Evaluation in Pulmonary Fibrosis
Acronym: FIBROMET
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Ceinge - Biotecnologie Avanzate s.c. a r.l. (Unknown)
Responsible Party: Principal Investigator, Andrea Bianco, Full Professor, University of Campania Luigi Vanvitelli
Other Study IDs: 7721
Record Dates: First submitted 2025-04-25; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Pulmonary Fibrosis
Keywords: Metabolomic; Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pulmonary Fibrosis patients
  Interventions: Diagnostic Test: Fatty acids measurement

INTERVENTIONS:
Diagnostic Test: Fatty acids measurement — Serum analysis for metabolomic biomarker identification

SUMMARY:
Pulmonary fibrosis (PF) are a heterogeneous group of interstitial lung diseases who may have a progressive phenotype often associated with loss of lung function, chronic respiratory symptoms, quality of life limitation as well significant morbidity and mortality. The identification of reliable biomarkers able to help in early diagnosis and predict disease progression are crucial for improving patient life. Although many biomarkers have been proposed, there is no consensus on reliable markers for IPF. Alterations in fatty acid (FA) metabolism have drawn increasing attention in the IPF pathogenesis, but there is no consensus on the specific FA changes. Alterations in FA composition have been shown to promote pro-fibrotic traits in epithelial cells, fibroblasts, and myofibroblasts. However, while specific fatty acid (FA) alterations have been identified in the serum of IPF patients, no consensus exists on the exact changes for individual FAs

ELIGIBILITY:
Inclusion Criteria:

* Confirmed IPF diagnosis based on the 2018 ATS/ERS/JRS/ALAT guidelines [PMID: 30168753] or other fibrotising ILDs within the past five years,
* Age ≥ 40 years, 3) ability to provide informed consent.

Exclusion Criteria:

* A current diagnosis of asthma or chronic obstructive pulmonary disease (COPD), 2) an acute PF exacerbation within the past three months.
* Use of medications who may alter metabolomic biomarkers, ex. statins.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with a diagnosis of IPF or other fibrotising interstitial lung disease within 5 years
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2025-01-18 (Actual)

PRIMARY OUTCOMES:
Fatty acids measurement | six months

CONTACTS AND LOCATIONS:
Locations (1):
- UOC Clinica Pneumologica L Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/99/NCT06974799/Prot_SAP_000.pdf